CLINICAL TRIAL: NCT04245475
Title: Water-friendly Virtual Reality and Brief Thermal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Hunter Hoffman, Research Scientist: Radiology, Psychology, Engineering, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00007801; R01GM042725 (NIH)
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Pain, Acute
Keywords: pain control
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Within subjects crossover design, VR treatment order randomized (some participants receive Low Tech VR + High Tech VR, some participants receive High Tech VR + Low Tech VR) and some participants receive No VR in a side study to test the assumptions of our QST testing pain paradigm.
  1. No Virtual Reality (no treatment control side data to test QST paradigm assumptions).
  2. Low Tech/passive Virtual Reality for 1st pain stimulus+High Tech for 2nd pain stimulus
  3. High Tech/interactive VR for 1st pain stimulus +Low Tech for 2nd pain stimulus.
Who Masked: Outcomes Assessor
Masking Description: Some of the instructions for the outcome measure will be presented to the participants via a computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No treatment, side study to test the assumptions of our quantitative sensory testing pain paradigm
- Low Tech/passive Virtual Reality first (Active Comparator): Low Tech VR first brief test phase thermal stimulus + High Tech VR during a second test phase pain stimulus
  Interventions: Behavioral: Virtual Reality psychological pain reduction
- High Tech/interactive Virtual Reality first (Experimental): High Tech/Interactive VR during first brief test phase thermal stimulus + Low Tech VR during a second brief thermal stimulus.
  Interventions: Behavioral: Virtual Reality psychological pain reduction

INTERVENTIONS:
Behavioral: Virtual Reality psychological pain reduction — attention distraction
  Arms: High Tech/interactive Virtual Reality first; Low Tech/passive Virtual Reality first

SUMMARY:
Using immersive virtual reality as a form of pain distraction during a brief "painful but tolerable" temperature.

DETAILED DESCRIPTION:
This study will use Quantitative Sensory Testing (computer-controlled brief 10 second thermal pain stimuli) in healthy college students.

The primary aim is to conduct a randomized, controlled study with healthy volunteers to explore whether interacting with virtual objects in VR via a high tech interactive VR system makes VR significantly more effective/powerful compared to a less immersive passive VR system, vs. No VR, for reducing pain during quantitative sensory testing.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a course at the University of Washington Psychology Dept., participating in the UW Psychology subject pool
* Able to read, write and comprehend English
* Able to complete study measures
* Willing to follow our UW approved instructions
* 18 years of age or older

Exclusion Criteria:

* People how have already previously participated in this same study (e.g., last quarter) are not eligible to participate again.
* Not enrolled in a course at the University of Washington Psychology Dept., participating in the UW Psychology subject pool
* Not be able to read, write and comprehend English
* Younger than 18 years of age.
* Not capable of completing measures
* Not capable of indicating pain intensity,
* Not capable of filling out study measures,
* Extreme susceptibility to motion sickness,
* Seizure history,
* Unusual sensitivity or lack of sensitivity to pain,
* Sensitive skin,
* sensitive feet,
* migraines,
* Diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
participants rating of "worst pain " | immediately after each single 10 second test phase quantitative sensory test stimulus during a single visit
  using a single graphic rating scale, 0 = no pain, 10 = excruciating pain

SECONDARY OUTCOMES:
participants rating of "time spent thinking about pain" | immediately after each single 10 second quantitative sensory test stimulus during a single visit
  using a single graphic rating scale, 0 = none of the time, 10 = all of the time
participants rating of "pain unpleasantness " | immediately after each single 10 second quantitative sensory test stimulus during a single visit
  using a single graphic rating scale, 0 = no pain, 10 = excruciating pain

OTHER OUTCOMES:
participants rating of "fun" | immediately after each single 10 second quantitative sensory test stimulus during a single visit
  using a single graphic rating scale, 0 = no fun, 10 = extremely fun.

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Hoffman, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington (public not eligible for participation), Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Hoffman HG. Interacting with virtual objects via embodied avatar hands reduces pain intensity and diverts attention. Sci Rep. 2021 May 21;11(1):10672. doi: 10.1038/s41598-021-89526-4. PMID 34021173